CLINICAL TRIAL: NCT00422318
Title: Hyperuricemia and the Effects of the Uricosuric Agents Benzbromarone in Patients With Chronic Heart Failure
Brief Title: Treatment of Hyperuricemia in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tottori University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #345
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Heart Failure; Hyperuricemia
Keywords: Heart Failure; Insulin; Metabolism; Pharmacology; Uric Acid
MeSH Terms: conditions — Heart Failure; Hyperuricemia; Insulin Resistance | interventions — Benzbromarone; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Benzbromarone (drug)

SUMMARY:
The study aims to assess (I) the contribution of UA itself to the CHF pathophysiology and (II) to test the effect of lowering UA by uricosuric treatment in CHF.

DETAILED DESCRIPTION:
Hyperuricemia is often observed in patients with congestive heart failure (CHF). It has been reported that hyperuricemia is related to exercise capacity, inflammation markers and diastolic dysfunction in such patients. In addition, hyperuricemia in CHF relates to both symptomatic status (i.e. morbidity) as well as impaired prognosis (i.e. mortality). Hyperuricemia is likely to play an important role in the pathophysiology of CHF. Up-regulation of xanthine oxidase (XO) activity in CHF has been shown to contribute to higher uric acid (UA) in CHF and the therapeutic concept of XO inhibition has shown beneficial effects in a number of surrogate markers in these patients. The XO inhibition accounts for substantial decrease in oxygen radical load, the latter is discussed as the main benefit of XO inhibition treatment in hyperuricemic patients. However, whether high uric acid itself is important or merely a marker of XO activity (and hence of increased radical accumulation) is currently under discussion. Therefore, this study aims to assess (I) the contribution of UA itself to the CHF pathophysiology and (II) to test the effect of lowering UA by uricosuric treatment in CHF.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure
* hyperuricemia

Exclusion Criteria:

* renal dysfunction (Cr > 2.0 mg/dl)
* under treatment with anti-diabetic agents

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-01; Study Completion 2005-12

PRIMARY OUTCOMES:
parameters of echocardiography at 16 weeks
BNP levels at 16 weeks

SECONDARY OUTCOMES:
parameters of glucose metabolism at 16 weeks
Parameters of lipid metabolism at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhide Ogino, MD, Principal Investigator — Tottori University Hospital
Locations (1):
- Tottori University Hospital, Yonago, Japan

REFERENCES:
- [Derived] Ogino K, Kato M, Furuse Y, Kinugasa Y, Ishida K, Osaki S, Kinugawa T, Igawa O, Hisatome I, Shigemasa C, Anker SD, Doehner W. Uric acid-lowering treatment with benzbromarone in patients with heart failure: a double-blind placebo-controlled crossover preliminary study. Circ Heart Fail. 2010 Jan;3(1):73-81. doi: 10.1161/CIRCHEARTFAILURE.109.868604. Epub 2009 Nov 20. PMID 19933411